CLINICAL TRIAL: NCT07380854
Title: Thyroid Hormone Replacement After Coronary Artery Bypass Grafting for Patients With Subclinical Hypothyroidism
Acronym: RepleniSH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Min Joo Kim, Professor of Internal Medicine, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-B-2110-717-003
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Subclinical Hypothyroidism
Keywords: subclinical hypothyroidism; coronary artery bypass grafting; thyroid hormones; levothyroxine
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LT4 group (Experimental): Participants in this group will receive levothyroxine
  Interventions: Drug: levothyroxine
- Control group (No Intervention): Participants in this group will not receive levothyroxine

INTERVENTIONS:
Drug: levothyroxine — Intervention description: Participants assigned to the LT4 group will begin receiving levothyroxine the day before CABG. The initial dose is 25 μg once daily, or 12.5 μg for participants weighing less than 60 kg. The dose will then be adjusted based on thyroid function test results to achieve target TSH levels of 0.4-2.0 μIU/mL.
  Arms: LT4 group

SUMMARY:
The goal of this clinical trial is to find out whether levothyroxine reduces complications and improves the prognosis of patients with subclinical hypothyroidism (SCH) undergoing coronary artery bypass grafting (CABG).

The main questions this study aims to answer are:

• Does levothyroxine reduce major adverse cardiovascular events (MACE), including cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and new arrhythmias, in SCH patients undergoing CABG? Researchers will compare patients who take levothyroxine with those who do not.

Participants will:

* Be randomly assigned to either receive levothyroxine or not
* Start the medication one day before surgery if assigned to the treatment group.
* Have regular follow-up visits to check thyroid function and cardiovascular events for up to five years after surgery.

ELIGIBILITY:
Eligibility Criteria

* Adults aged 19 to 90 years.
* Patients scheduled to undergo coronary artery bypass graft (CABG) surgery.
* Subclinical hypothyroidism (SCH), defined as a normal free thyroxine (free T4) level and a thyroid-stimulating hormone (TSH) level greater than 4 μIU/mL, based on testing performed within 31 days prior to surgery.

Exclusion Criteria:

* Patients who underwent repeat or emergency CABG surgery
* Use of LT4 within the previous 4 weeks
* Use of antithyroid drug use (propylthiouracil, methimazole, or carbimazole) within the previous 3 months
* Severe comorbid conditions with a life expectancy of less than 1 year (e.g. advanced malignancy)

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2022-02-27 (Actual); Primary Completion 2032-02-26 (Estimated); Study Completion 2037-02-26 (Estimated)

PRIMARY OUTCOMES:
A composite of MACE within 4months after surgery | within 4months after surgery
  A composite of major adverse cardiovascular events (MACE), including cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and the occurrence of new arrhythmias assessed within 4 months after CABG.

SECONDARY OUTCOMES:
Number of participants who experience cardiovascular death within 4 months after surgery | within 4months after surgery
  Number of participants who experience cardiovascular death within 4 months after CABG
Number of participants who experience nonfatal myocardial infarction within 4 months after surgery | within 4months after surgery
  Number of participants who experience nonfatal myocardial infarction within 4 months after CABG
Number of participants who experience nonfatal stroke within 4 months after surgery | within 4months after surgery
  Number of participants who experience nonfatal stroke within 4 months after CABG
Number of participants who experience new arrhythmia within 4 months after surgery | within 4months after surgery
  Number of participants who experience new arrhythmia within 4 months after CABG
A composite of MACE within 1 year after surgery | within 1 year after surgery
  A composite of major adverse cardiovascular events (MACE), including cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and the occurrence of new arrhythmias assessed within 1year after CABG
A composite of MACE within 5 year after surgery | within 5 years after surgery
  A composite of major adverse cardiovascular events (MACE), including cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and the occurrence of new arrhythmias assessed within 5 years after CABG
All-cause mortality within 5 years after surgery | within 5 years after surgery
  All-cause mortality within 5 years after surgery
Change in LVEF from baseline to 1 year after surgery | From baseline to 1 year after surgery
  Left ventricular ejection fraction (LVEF) will be measured using transthoracic echocardiography at baseline (pre-operative) and at 1 year post-operatively. The outcome will be reported as the mean change in LVEF (%) from baseline to 1 year.
Change in LV EDD from baseline to 1 year after surgery | From baseline to 1 year after surgery
  Left ventricular end-diastolic diameter (LVEDD) will be measured using transthoracic echocardiography at baseline (pre-operative) and at 1 year post-operatively. The outcome will be reported as the mean change in LVEDD (%) from baseline to 1 year.
Change in LV ESD from baseline to 1 year after surgery | From baseline to 1 year after surgery
  Left ventricular end-systolic diameter (LV ESD) will be measured using transthoracic echocardiography at baseline (pre-operative) and at 1 year post-operatively. The outcome will be reported as the mean change in LV ESD (%) from baseline to 1 year.
Change in LVMI from baseline to 1 year after surgery | From baseline to 1 year after surgery
  Left ventricular mass index (LVMI) will be measured using transthoracic echocardiography at baseline (pre-operative) and at 1 year post-operatively. The outcome will be reported as the mean change in LVMI (%) from baseline to 1 year.
Change in LAMI from baseline to 1 year after surgery | From baseline to 1 year after surgery
  Left atrial volume index (LAMI) will be measured using transthoracic echocardiography at baseline (pre-operative) and at 1 year post-operatively. The outcome will be reported as the mean change in LAMI (%) from baseline to 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No